CLINICAL TRIAL: NCT01762436
Title: A Randomized Controlled Study: Effects of Bisoprolol and Atenolol on Sympathetic Nervous Activity and Central Aortic Pressure in Patients With Essential Hypertension
Brief Title: Effects of Bisoprolol and Atenolol on Sympathetic Nervous Activity and Central Aortic Pressure in Patients With Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Weijun Zhou, Associate Profeesor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Betablocker on CAP and BRS
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Untreated Essential Hypertension
MeSH Terms: interventions — Bisoprolol; Atenolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bisoprolol (Experimental): initially received 5 mg of bisoprolol (Concor®, Merck Serono, Darmstadt, Germany) once daily. The heart rate was assessed every two weeks. If the RHR was ≤65 bpm, a 2-week maintenance treatment was added during the final visit. If the target RHR was not achieved, the dose was changed as recommended in the study protocol. The maximal dose was 10 mg Qd for bisoprolol. The longest treatment period was 8 weeks. If the patient's RHR did not reach below 65 bpm at week 6, the treatment was ended at week 8.
  Interventions: Drug: bisoprolol
- atenolol (Active Comparator): initially received 50 mg atenolol (Beijing Double-Crane Pharmaceutical Co., Ltd, Beijing, China) once daily. The heart rate was assessed every two weeks. If the RHR was ≤65 bpm, a 2-week maintenance treatment was added during the final visit. If the target RHR was not achieved, the dose was changed as recommended in the study protocol. The maximal dose was 100 mg Qd for atenolol. The longest treatment period was 8 weeks. If the patient's RHR did not reach below 65 bpm at week 6, the treatment was ended at week 8.
  Interventions: Drug: atenolol

INTERVENTIONS:
Drug: bisoprolol
  Arms: bisoprolol
Drug: atenolol
  Arms: atenolol

SUMMARY:
β-blockers (BBs) with different pharmacological properties may have heterogeneous effects on sympathetic nervous activity (SNA) and central aortic pressure (CAP), which are independent cardiovascular factors for hypertension. Hence, we analyzed the effects of bisoprolol and atenolol on SNA and CAP in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* 25~65 years old
* untreated essential hypertension
* SBP 140-160mmHg & DBP 90-100mmHg
* Sinus rhythm
* Resting heart rate >70bpm
* Can give written informed consent

Exclusion Criteria:

* Atrial Fibrillation (AF)/ Sick Sinus Syndrome (SSS)/ atrioventricular block 2-3 grade(AVBⅡ-Ⅲ) without pacemaker
* Bradyarrhythmia/ hypotensive
* Unstable Angina Pectoris (UAP)/AMI/ HF (NYHA class III - IV)
* Uncontrolled diabetes mellitus (DM)
* Bronchial asthma
* Gastro-intestinal ulcer or skin ulcer
* Liver dysfunction/ renal impairment
* Treated with CCB (Calcium antagonists) ( except amlodipine) or other beta blocker.
* Glaucoma
* Known allergic/ intolerance to beta blocker
* Pregnant or lactating women
* Participation in another clinical study within the last 3 months
* Legal incapacity or limited legal capacity

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
baroreflex sensitivity | 4~8 weeks
  After 2-week maintenance treatment when the RHR was ≤65 bpm or at 8-week final visit
central aortic pressure | 4~8 weeks
  After 2-week maintenance treatment when the RHR was ≤65 bpm or at 8-week final visit

SECONDARY OUTCOMES:
heart rate variability | 4~8 weeks
  After 2-week maintenance treatment when the RHR was ≤65 bpm or at 8-week final visit
peripheral blood pressure | 4-8 weeks
  After 2-week maintenance treatment when the RHR was ≤65 bpm or at 8-week final visit
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 4-8 weeks
  After 2-week maintenance treatment when the RHR was ≤65 bpm or at 8-week final visit

CONTACTS AND LOCATIONS:
Locations (1):
- State Key Laboratory of Medical Genomics, Shanghai Key Laboratory of Hypertension and Department of Hypertension, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhou WJ, Wang RY, Li Y, Chen DR, Chen EZ, Zhu DL, Gao PJ. A randomized controlled study on the effects of bisoprolol and atenolol on sympathetic nervous activity and central aortic pressure in patients with essential hypertension. PLoS One. 2013 Sep 10;8(9):e72102. doi: 10.1371/journal.pone.0072102. eCollection 2013. PMID 24039738